CLINICAL TRIAL: NCT06504628
Title: CHUtes Chez Les Personnes Agées traitées Pour Cancer Dans Les HOpitaUx Normands : repérage et Prévention
Brief Title: Falls Among the Older Patients Treated for Cancer in Normandy's Outclinics: Screening and Prevention
Acronym: CHUPACHOUP
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00979-38
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-09

CONDITIONS: Aged Patients Treated for Cancer in Outclinics
Keywords: aged; outpatients; cancer; accidental falls
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low risk for fall subgroup: according to Manuel Montero-Odasso M, Nathalie van der Velde, Finbarr C Martin, Mirko Petrovic, Maw Pin Tan, Jesper Ryg, et al. World guidelines for falls prevention and management for older adults: a global initiative. Age and Ageing, Volume 51, Issue 9, September 2022
  Interventions: Diagnostic Test: screening risk for falling and identifiy the risk level low-intermediate-high
- intermediate risk for fall subgroup: according to Manuel Montero-Odasso M, Nathalie van der Velde, Finbarr C Martin, Mirko Petrovic, Maw Pin Tan, Jesper Ryg, et al. World guidelines for falls prevention and management for older adults: a global initiative. Age and Ageing, Volume 51, Issue 9, September 2022
  Interventions: Diagnostic Test: screening risk for falling and identifiy the risk level low-intermediate-high
- high risk for fall subgroup: according to Manuel Montero-Odasso M, Nathalie van der Velde, Finbarr C Martin, Mirko Petrovic, Maw Pin Tan, Jesper Ryg, et al. World guidelines for falls prevention and management for older adults: a global initiative. Age and Ageing, Volume 51, Issue 9, September 2022.
  Those patients will be contacted 3 mnths after inclusion for follow-up assessment
  Interventions: Diagnostic Test: screening risk for falling and identifiy the risk level low-intermediate-high; Diagnostic Test: 3 mnth-follow-up

INTERVENTIONS:
Diagnostic Test: screening risk for falling and identifiy the risk level low-intermediate-high — 3 key questions: Any posiitve answer to a) Has fallen in the past year? b) Feels unsteady when standing or walking? or c) Worries about falling? prompts to "fall severity" step.
  if "no" at the three questions= low level of fall-risk Fall severity: fall with injuires, laying on the ground with no capacity to get up, or a visit to emergency room, or loss of conscienciousness/suspected syncope. or Frailty (Clinical Frailty Scale)= if positive, high risk otherwise, 4 meter-walk test: if =<0.8m/sec= intermediate risk if >0.8m/sec=intermediate risk
  Other Names: prevention by handing over a leeflet listing recommendations to patients and general practitionners
Diagnostic Test: 3 mnth-follow-up — patient's phone call, and data collected from electronic medical record
  Groups: high risk for fall subgroup

SUMMARY:
The French Plan National AntiChute (published on February 21, 2022) and international recommendations on falls prevention (Age Ageing,September 2022) recommend identifying the risk of falling in people aged 65 and over, at least once a year during a follow-up consultation. The presence of chronic illness such as cancer increases the risk for falling. Recommendations suggest targeted preventive interventions according to the risk level, and early reassessment at 3 months in case of high risk.

This study consists of a cross-sectional survey conducted during a week dedicated to patient safety (September 16-20, 2024), to identify the prevalence of patients at high risk for falling, requiring enhanced care. The relation between high risk for falling and social and oncological characteristics will be studied. A 3-month telephone follow-up will identify any obstacles to implementing the recommendations in this high-risk group.

This multicenter cross-sectional prospective study is exploratory.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 or over
* undergoing treatment for cancer or hematological malignancy (oral or injectable systemic treatment, radiotherapy)
* covered by health insurance
* having read the information document and no objection
* French-speaking
* Autonomous ( with occasional assistance with instrumental daily activities),

Exclusion Criteria:

* refusal to participate
* unable to communicate
* dependent (requiring geriatric care)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 and over treated for cancer or haematological malignancy in public and private outclinics -hospitals in Normandy
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
prevalence of each of the three levels of fall-risk | Day 1
  describe the distribution of patients in mild, intermediate and high risk for falling

SECONDARY OUTCOMES:
look for association between high-risk categorization and rural place of residence, gender, age bracket (65-74 and 75 and over), investigating center, type of cancer (location). | Day 1
Describe the rate of high-risk patients who will have benefited from (full or partial) implementation of recommended interventions according to 3-month follow-up. | 3 mnths
among high-risk patients followed up at 3 months, look for an association between the absence ofimplementation of recommendations and social, medical characteristics and motive | 3 mnths
describe the Average number of STOPPFALL medications per patient. Rate of patients with at least one oncologydrug listed as a fall risk (CIPN), in the 3 fall risk categories | Day 1

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Caen UH, Caen, Normandy
  - Centre de radiothérapie de la Baie, Avranches
  - Centre de radiothérapie Maurice Tubiana/Polyclinique Parc, Caen
  - CLCC François Baclesse, Caen
  - Centre Hospitalier Public du Cotentin, Cherbourg
  - Centre Hospitalier Evreux-VErnon, Évreux
  - Hôpital Privé de l Estuaire, Le Havre
  - Centre Hospitalier Robert Bisson, Lisieux
  - Becquerel Cancer CEnter, Rouen
  - CHU de Rouen Charles Nicolle, Rouen